CLINICAL TRIAL: NCT04783480
Title: Can Birthly, an Online Childbirth Education Platform, Reduce Pregnancy-related Anxiety Compared to Usual Care: An RCT
Brief Title: Can Birthly, an Online Childbirth Education Platform, Reduce Pregnancy-related Anxiety Compared to Usual Care
Acronym: Birthly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 848373
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy, High Risk
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Birthly plus standard of care (Active Comparator): Women will receive a code to sign up for childbirth education classes through the Birthly platform. They will also participate in childbirth education at their own discretion.
  Interventions: Other: Birthly
- Standard of Care (Placebo Comparator): Women will not receive a code for the 3 Birthly courses. They will participate in childbirth education at their own discretion.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Birthly — Women will receive a code to sign up for 3 free interactive childbirth education classes through the Birthly platform. They will be enrolled in 3 courses: Prenatal Education, Childcare and Breastfeeding. They will be encouraged to complete all courses prior to 36 weeks gestational age.
  Arms: Birthly plus standard of care
Other: Standard of care — Subjects will participate in childbirth education at their own discretion.
  Arms: Standard of Care

SUMMARY:
A pilot randomized, controlled trial comparing Birthly, (an online platform for live group prenatal classes taught by childbirth educators, nurses, and lactation consultants) plus standard prenatal care versus standard prenatal care alone among women with high risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* Willing and stable to give consent
* English-speaking
* Have access to high-speed internet available on a computer or mobile device
* Nulliparous women have a confirmed single, live intrauterine gestation and are <20 weeks gestational age at their prenatal visit
* Women without indications for a scheduled cesarean delivery at the time of their index prenatal visit
* Women who have a high-risk pregnancy, as defined by all maternal conditions including hypertension, diabetes, auto-immune disorders, seizure disorder, substance use, etc
* Agree to participation in Birthly
* Obtaining prenatal care in the University of Pennsylvania Health System

Exclusion Criteria:

* Women who do not speak at least conversational English
* Women without internet access
* Multiparous women
* Women receiving group prenatal care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in PrAS score | time of enrollment to 34-40 weeks gestation
  To determine if access to an online comprehensive platform for prenatal education and childbirth courses decreases pregnancy anxiety as measured by the Pregnancy-Related Anxiety Scale (PrAS) in nulliparous women with high risk pregnancies compared to usual prenatal care. The primary study endpoint will be a 15% reduction in PrAS score from 64 to 55 with a SD of 15.22.

SECONDARY OUTCOMES:
Difference in healthcare utilization | time of enrollment through 6-week postpartum
  Measured by the number of unscheduled visits to the obstetrical triage unit or ED, urgent office visits, and triage telephone encounters during pregnancy and in the 6-week postpartum period
Difference in Edinburgh Postnatal Depression Scale | one-time score at 4-6 weeks postpartum
  The scoring scale is 1 to 30, with a higher score indicating a worse outcome
Difference in intention to breastfeed | at 34 to 40 weeks gestational age
  Intention to breastfeed prior to delivery
Difference in breastfeeding rates at discharge after delivery | time of discharge from hospital after delivery
Difference in breastfeeding rates postpartum | 4-6 weeks postpartum
Difference in contraceptive uptake at discharge from hospital | at time of discharge from hospital after delivery, on average 1-3 days postpartum
Difference in contraceptive uptake postpartum | 4-6 weeks postpartum
Mode of delivery | delivery
Number of participants with hypertensive disorders of pregnancy | delivery through 4-6 weeks postpartum
Number of participants with maternal readmission | delivery through 4-6 weeks postpartum
Number of participants who have Preterm birth | Time of delivery
Difference in APGAR scores | Time of birth
Number of infants with a need for neonatal respiratory support outside the delivery room | Time of birth
Number of infants with a NICU admission | Time of birth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zafman KB, Riegel ML, Levine LD, Hamm RF. An interactive childbirth education platform to improve pregnancy-related anxiety: a randomized trial. Am J Obstet Gynecol. 2023 Jul;229(1):67.e1-67.e9. doi: 10.1016/j.ajog.2023.04.007. Epub 2023 Apr 11. PMID 37054807